CLINICAL TRIAL: NCT00651833
Title: An Open-Label, Non-Randomized, Multicenter, Three-Stage, Phase 2 Study of S-1 in Combination With Cisplatin as 1st Line Therapy for Patients With Advanced Non-Small Cell Lung Cancer (Stage IIIB/Stage IV)
Brief Title: Phase 2 Study of S-1 in Combination With Cisplatin as 1st Line Therapy in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry); United BioSource, LLC (Industry)
Responsible Party: Fabio Benedetti, M.D., Chief Medical Officer, Taiho Pharma USA, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1202; NCT00227578 (obsolete NCT alias)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All patients will receive S-1 orally at a dose of 25 mg/m2 twice daily (BID) for 14 days followed by a 1-week recovery period, repeated every 3 weeks. Patient will also receive cisplatin, 75 mg/m2 as a 1- to 3-hour infusion on Day 1 of each cycle.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — All patients will receive S-1 orally at a dose of 25 mg/m2 twice daily (BID) for 14 days followed by a 1-week recovery period, repeated every 3 weeks. The study may go to the third stage only if 7/31 (23%) or more patients have achieved a confirmed response (CR or PR) in stages 1 and 2 combined.

SUMMARY:
The purpose of this study is to determine whether S-1 in combination with Cisplatin is effective as 1st line therapy in slowing tumor activity in patients with advanced non-small cell lung cancer. The study is also looking at the safety of S-1.

DETAILED DESCRIPTION:
Advanced non-small cell lung cancer is relatively unresponsive to chemotherapy. This is true for the nucleoside analogue gemcitabine, with a response rate of approximately 10%, as well as for 5-fluorouracil (5-FU). Even when gemcitabine is combined with other chemotherapeutic drugs or biological agents, the overall tumor response rate remains basically unchanged. S-1 is a new generation oral fluoropyrimidine that combines Tegafur (5-fluoro-1-(tetrahydro-2-furanyl)-2,4(1H,3H)-pyrimidinedione [FT]), an oral prodrug of 5-FU, with two modulators, Gimeracil (5-chloro-2,4-dihydroxypyridine [CDHP]), which inhibits 5-FU degradation by dihydropyrimidine dehydrogenase (DPD) inhibition, and Oteracil potassium (Oxo), which inhibits 5-FU phosphorylation in the digestive tract. This combination of 3 compounds is designed to achieve enhanced antitumor activity while decreasing gastrointestinal toxicity.

This is an open-label, multicenter, single-arm, 3-stage, Phase 2 study evaluating the efficacy and safety of S-1 in combination with cisplatin as 1st line therapy for patients with advanced NSCLC. The 3 stages of this study correspond to a run-in tolerability stage (stage 1), futility stage (stage 2), and decision stage (stage 3). The run-in tolerability stage will be conducted to assess any additional toxicity associated with a more frequent schedule of administration of cisplatin (75 mg/m2 every 3 weeks) compared with the dosing regimen established in a prior Phase I study in patients with advanced gastric cancer (75 mg/m2 every 4 weeks). The futility stage (stage 2) will be conducted to ensure that this treatment combination is sufficiently efficacious to expose a sufficient number of patients to be able to make a decision (stage 3) on whether this combination treatment warrants further evaluation in future studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Has given written informed consent. 2. Patients with histologically and/or cytologically proven unresectable NSCLC stage IIIB with pleural effusion or pericardial effusion, or stage IV (mixed forms with small cell lung cancer are excluded).

  3. Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, ie, has at least one measurable lesion. A measurable lesion is one that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral Computed Tomography (CT) scan.

  4. Is able to take medications orally. 5. Is ≥ 18 years of age. 6. Has an ECOG performance status 0 or 1. 7. Has adequate organ function as defined by the following criteria:
  1. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN; if liver function abnormalities are due to underlying liver metastasis AST (SGOT) and ALT (SGPT) ≤ 5 x ULN.
  2. Total serum bilirubin of ≤ 1.5 x ULN.
  3. Absolute granulocyte count of ≥ 1,500/mm3.
  4. Platelet count ≥ 100,000/mm3.
  5. Hemoglobin of ≥ 9.0 g/dL.
  6. Calculated creatinine clearance (CrCl) ≥ 60 mL/minute (Cockcroft-Gault formula).

     8. Is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

     Exclusion Criteria:
* 1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

  1. Any prior cytotoxic chemotherapy except for adjuvant or neo-adjuvant therapy for NSCLC beyond 12 months.
  2. Any radiation therapy to a target lesion unless there was evidence of PD after radiotherapy (and this target lesion must not be the only site of measurable disease).
  3. Radiotherapy within the prior 2 weeks.
  4. Adjuvant or neo-adjuvant therapy within the past 12 months.
  5. Prior cisplatin as neo-adjuvant and/or adjuvant chemotherapy with cumulative dose > 300 mg/m2.
  6. Any investigational agent, either concurrently or within the past 30 days.
  7. Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study.

     2. Has a serious illness or medical condition(s) including, but not limited to, the following:

  <!-- -->

  1. Other active malignancies.
  2. Symptomatic brain metastasis not controlled by corticosteroids.
  3. Leptomeningeal metastasis.
  4. Known neuropathy Grade 2 or higher.
  5. Myocardial infarction within the last 6 months, severe/unstable angina, congestive heart failure New York Heart Association (NYHA) class III or IV.
  6. Chronic nausea, vomiting, and/or diarrhea.
  7. Psychiatric disorder that may interfere with consent and/or protocol compliance.
  8. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
  9. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.

     3. Is receiving concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

  <!-- -->

  1. Sorivudine, uracil, cimetidine, folinic acid, and dipyridamole (may enhance S-1 activity).
  2. Allopurinol (may diminish S-1 activity).
  3. Phenytoin (S-1 may enhance phenytoin activity).
  4. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 activity).4. Is receiving concomitant treatment with drugs interacting with cisplatin. The following drugs are prohibited because there may be an interaction with cisplatin:

  <!-- -->

  1. Phenytoin (cisplatin may diminish phenytoin activity).
  2. Aminoglycosides (should be avoided within 8 days after cisplatin administration).

     5. Is a pregnant or lactating female. 6. Has known hypersensitivity to cisplatin. 7. With reproductive potential and refuses to use an adequate means of contraception (including male patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-02; Primary Completion 2006-10 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall tumor response rate (ORR - the proportion of patients with objective evidence of PR or CR) | Each cycle will last 21 days (14 days treatment, 7 days recovery) for a max of 6 cycles. Tumor assessments will be obtained at baseline and at the end of every even cycle.

SECONDARY OUTCOMES:
To evaluate the safety profile of S-1 | AEs will be reported through follow-up (30 days after the last dose of study medication); blood/urine will be collected at baseline ; Days 8 and 15; w/in 24 hrs prior to study drug on Day 1 of each cycle after Cycle 1; at the end of study treatment.
To evaluate the duration of response (DR), and progression-free survival (PFS) | Each cycle will last 21 days (14 days treatment, 7 days recovery) for a max of 6 cycles. Following discont'n of treatment , pts will be followed for survival status every 2 mos following PD for up to 6 mos.
To investigate the relationship of S-1 plasma levels (components and metabolites) with safety and efficacy parameters | Each cycle will last 21 days (14 days treatment, 7 days recovery) for a max of 6 cycles. Blood samples to be obtained 1.5 ± 0.5 h, 5 ± 1 h, 7 ± 1 h postdose on Day 1 of Cycle 1 only.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Benedetti, MD, Study Director — Taiho Oncology, Inc.